CLINICAL TRIAL: NCT00809822
Title: NPB-01(Intravenous Immunoglobulin) Therapy for Patients With Bullous Pemphigoid Unresponsive to Corticosteroids: Randomized, Double-Blind, Placebo Control,Parallel Assignment Study(PhaseⅡ).
Brief Title: Clinical Trial of NPB-01 in Patients With Bullous Pemphigoid Unresponsive to Corticosteroids.
Acronym: NPB-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Nihon Pharmaceutical Co., Ltd, Clinical Development Department
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPB-01-06/E-01
Record Dates: First submitted 2008-12-11; First posted 2008-12-17 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Bullous Pemphigoid
Keywords: IVIG in pemphigoid; Patients with bullous pemphigoid unresponsive to corticosteroids
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Intravenous immunoglobulin
  Interventions: Drug: NPB-01
- 2 (Placebo Comparator): Physiological saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NPB-01 — Intravenous immunoglobulin
  Arms: 1
Drug: Placebo — Physiological saline
  Arms: 2

SUMMARY:
Patients diagnosed with bullous pemphigoid were confirmed based on the investigators national diagnostic criteria. Patients who meet all inclusion criteria and conflict the exclusion criteria will receive NPB-01(intravenous immunoglobulin) 400mg/kg/day for five consecutive days or Placebo(physiological saline). Subsequently, efficacy of NPB-01 for therapy of bullous pemphigoid will evaluate using pemphigoid activity score involving skin lesion area and Number of new blisters.

As a safety endpoint, the safety of NPB-01 will be investigated the occurrence of adverse events by 57 days after the start of the study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with corticosteroids over 20mg/day(Prednisolone) at informed consent.
2. Patients with continued treatment for bullous pemphigoid without add or change the treatment after informed consent.
3. Patients who pemphigoid activity score is score1 and more before study medication received.
4. Patients who symptom is not improve before study medication received.
5. Patients with twenty years old at informed consent.
6. Patients with hospitalization during five consecutive days of study medication.

Exclusion Criteria:

1. Patients treated with plasmapheresis at 28 days before informed consent.
2. Patients treated with corticosteroids pulse therapy(methylprednisolone over 0.5g/day) at 14 days before informed consent.
3. Patients treated with intravenous immunoglobulin at 56 days before informed consent.
4. Patients who receive or adjust in increments immunosuppressants at 14 days before informed consent.
5. Patients with malignancy or a history of this disease.
6. Patients with history of shock for NPB-01.
7. Patients with history of hypersensitivity for NPB-01.
8. Patients with IgA deficiency.
9. Patients with impaired liver function.
10. Patients with impaired renal function.
11. Patients with cerebro- or cardiovascular disorders.
12. Patients with high risk of thromboembolism.
13. Patients with hemolytic/hemorrhagic anemia.
14. Patients with decreased cardiac function.
15. Patients with decreased platelet.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Skin lesion area (%), Number of new blisters/day, Pemphigoid Activity Score, Pemphigus Disease Area Index(PDAI), anti-BP180 and -BP230 antibody titers, Steroid dose, Time to escape from the protocol and its ratio | 57 days

CONTACTS AND LOCATIONS:
Locations (1):
- Osaka, Japan